CLINICAL TRIAL: NCT00822159
Title: Prospective Multicenter Cohort Study to Evaluate the Influence of Bone Strength Measured by DensiProbe Hip on Bone Related Fixation Failure in Patients With Hip Fractures Undergoing DHS Surgical Treatment.
Brief Title: Influence of Bone Strength Measured by DensiProbe on Bone Related Fixation Failure
Acronym: Densiprobe
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis showed statistically significant results
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Densiprobe-08
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Femoral Fractures; Hip Fractures; Osteoporosis; Bone Density
Keywords: Fixation failure; Bone strength; DensiProbe
MeSH Terms: conditions — Femoral Fractures; Hip Fractures; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: DensiProbe Hip — DensiProbe (CE marked) is a mechanical probe, which is used intra-operatively to assess mechanical stability of the trabecular bone in the proximal femur. It consists of a drill bit like tool and an electronic system for measuring the peak torque to break-away of trabecular bone in the femoral head. DensiProbe measurements are designed to be integrated in the DHS surgical procedure.

SUMMARY:
Hip fractures mostly occur in elderly people with low bone strength. Bone strength is determined by bone mineral density (BMD), bone turnover, microarchitectural and geometrical properties of the bone. Dual energy x-ray absorptiometry (DXA) is the standard technique to measure BMD. However, BMD just provides information regarding the quantity of mineral in bone, which is only one component of bone strength. To date there is no reliable method to assess bone strength in vivo. Therefore, a method to assess bone strength beyond BMD would provide additional information regarding the patients' risk of bone related fixation failure after fracture fixation.

DensiProbe is a new diagnostic device that was developed for intra-operative assessment of mechanical stability of the bone in the proximal femur. It consists of a drill bit like tool and an electronic system to measure the peak torque to break-away of trabecular bone in the femoral head of patients undergoing DHS surgical treatment. In a cadaver study comparing bone mineral density measured by quantitative computed tomography with bone strength measured by DensiProbe a high correlation between these two parameters could be shown. In a clinical pilot study a significant correlation between DensiProbe measurements and BMD measured by DXA at the femoral neck in patients with hip fractures could be shown. However, no perfect correlation was expected because DensiProbe measures bone strength, which is only partly caused by BMD.

Bone related fixation failure, such as secondary loss of reduction, is influenced by bone strength, bone mineral density, fracture type, fracture reduction and primary positioning of the implant. The predictive value of DensiProbe measurements for secondary loss of reduction needs to be investigated. If DensiProbe turned out to be an effective screening tool for patients with low bone strength that are on higher risk of the aforementioned complications these patients may in future benefit from alternative treatment methods (e.g. augmentation techniques) in order to reduce bone related fixation failure.

The primary aim of the present study is to investigate if bone strength measured by DensiProbeTM Hip (DensiProbe) is an independent factor to predict secondary loss of reduction (screw migration of 5 mm or more and / or telescoping of 10 mm or more) in patients with hip fractures after fracture fixation with DHS.

ELIGIBILITY:
Inclusion Criteria:

* Patients 50 years or older
* Patients with trochanteric or femoral neck fractures, classified as: AO 31-A1, AO 31-A2, AO 31-A3, AO 31-B1, AO 31-B2, AO 31-B3
* Patients undergoing fixation with DHS (135° aiming device, anti-rotational K-wire)
* Patients willing to participate in the study according to the clinical investigation plan
* Patients able to understand and read country national language at an elementary level
* Signed written informed consent by the patient or legal guardian

Exclusion Criteria:

* Bilateral hip fractures (at present or in the past)
* Open hip fracture
* Any previous surgical procedures of the hip (ipsilateral / contralateral)
* More than 7 days between injury and surgery
* Polytrauma (multiple injuries, whereof one or the combination of several injuries is life-threatening)
* Patients being pregnant or breast-feeding
* Pathologic fractures
* Active malignancy
* Psychiatric disorders that would preclude reliable assessment (e.g. severe depression)
* Drug or alcohol abuse
* Patients having participated in any other device or drug related clinical trial within the previous month

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Migration of the screw in relation to the femoral head of 5 mm or more and/or Telescoping (shortening of the femoral neck) of 10 mm or more | 3 months

SECONDARY OUTCOMES:
Rate of complications | 3 months
BMD values measured by DXA (contralateral hip) | Post OP
Parker mobility score | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Suhm, MD, Principal Investigator — Universitätsspital Basel
Locations (8):
- Austria (2):
  - Medizinische Universität, Innsbruck
  - Wilhelminenspital, Vienna
- Germany (3):
  - Medizinische Hochschule Hannover, Hanover
  - Friedrich-Schiller Universität, Jena
  - Universitätsklinikum Münster, Münster
- Twenteborg Ziekenhuis Almelo, Almelo, Netherlands
- Switzerland (2):
  - Universitätsspital, Basel, Canton of Basel-City
  - Stadtspital Triemli, Zurich

REFERENCES:
- See also: Related Info — http://www.aofoundation.org